CLINICAL TRIAL: NCT05836441
Title: A Multicenter, Randomized, Open, Parallel Controlled Clinical Study Evaluating the Efficacy and Safety of Improved Phototherapy in Patients With Vitiligo
Brief Title: Improved Phototherapy in Patients With Vitiligo
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: The First Affiliated Hospital with Nanjing Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NJmedical
Record Dates: First submitted 2023-04-17; First posted 2023-05-01 (Actual); Last update posted 2023-05-01 (Actual); Status verified 2023-04

CONDITIONS: Vitiligo
MeSH Terms: conditions — Vitiligo | interventions — Tacrolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- White spot irradiation group (Active Comparator): Exposure to white patches
  Interventions: Radiation: Exposure to white patches
- White spot edge irradiation group (Experimental): Exposure to edge of white patches and normal skin around white patches
  Interventions: Radiation: Exposure to edge of white patches and normal skin around white patches

INTERVENTIONS:
Radiation: Exposure to white patches — Exposure to white patches
  Other Names: Tacrolimus
  Arms: White spot irradiation group
Radiation: Exposure to edge of white patches and normal skin around white patches — Exposure to edge of white patches and normal skin around white patches
  Arms: White spot edge irradiation group

SUMMARY:
Vitiligo is a common acquired depigmentation skin and mucosal disease in dermatology, with or without white hair. Vitiligo with white hair is difficult to treat. Phototherapy and topical therapy are the first line treatment methods for vitiligo. The peripheral leukoplakia irradiation of phototherapy covers the central area of the leukoplakia and performs phototherapy on the edge of the leukoplakia and surrounding normal skin. This study aims to compare the efficacy and safety of peripheral leukoplakia ultraviolet family phototherapy and leukoplakia family combination in the treatment of vitiligo.

ELIGIBILITY:
Inclusion Criteria:

* ① Age: 5 years old and above

  * Gender: unlimited

    * Types of vitiligo: sporadic vitiligo, facial and neck vitiligo, mixed vitiligo, undetermined vitiligo

      * Vitiligo course: unlimited; ⑤ Vitiligo activity level: stable period; ⑥ At least one white spot meets the following four conditions simultaneously: Location: limited to the neck, trunk, and limbs (excluding hairless areas of hands and feet); There are no contraindications for the use of NB UVB phototherapy and topical tacrolimus; Area: 1cm2 < white spot area < 1% body surface area; The vellus hair in the white spot area is all white; ⑦ It is agreed to discontinue all forms of treatment that may change the study outcome during the study period, including western medicine, traditional Chinese medicine, traditional Chinese patent medicines and simple preparations, biological agents, etc., such as Dihydroketiazide, 8-M0P, osteotonic, angelica dahurica, etc; Willing and able to follow the visit and treatment plan.

Exclusion Criteria:

* ① Segmental vitiligo, generalized vitiligo, mucosal vitiligo, and acromegaly vitiligo;

  * Degree of vitiligo activity: progression, rapid progression

    * Kobner phenomenon or white spots located at the site of skin trauma, or other subjects requiring emergency intervention;

      * Subjects who are sensitive to or have contraindications to ultraviolet radiation (suffering from photosensitive diseases such as xeroderma pigmentosum, porphyria, Bloom syndrome, systemic lupus erythematosus, dysplastic nevus syndrome, dermatomyositis, etc.);

        * Subjects with a history of malignant tumors (including skin squamous cell carcinoma, melanoma or other skin and systemic malignant tumors);

          * Subjects with severe systemic diseases;

            * Subjects who are allergic to tacrolimus ointment or excipients in the ointment; ⑧ Subjects who have received oral or systemic medication (such as corticosteroids, cyclosporine, methotrexate, tacrolimus, etc.) aimed at controlling/improving vitiligo symptoms within 4 weeks prior to baseline, or who require systemic use of corticosteroids or immunosuppressants for other reasons;

              ⑨ Subjects who have received any optical therapy (including sunbathing) for vitiligo within 4 weeks prior to baseline;

              ⑩ Subjects who have received topical treatment aimed at controlling/improving vitiligo symptoms (such as glucocorticoids, calcineurin inhibitors, vitamin D3 derivatives, etc.) within 2 weeks prior to baseline.

              ⑪ Pregnant and lactating female subjects;

              ⑫ Subjects who are judged by researchers to be unable to implement treatment plans correctly;

              ⑬ Child subjects who cannot cooperate with phototherapy protective measures;

Min Age: 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 110 (Estimated)
Dates: Start 2022-01-01 (Actual); Primary Completion 2023-07-30 (Estimated); Study Completion 2023-12-30 (Estimated)

PRIMARY OUTCOMES:
percentage reduction in vitiligo area | week12 after intervention
  mean percentage reduction in vitiligo area from baseline to week 12

SECONDARY OUTCOMES:
percentage reduction of leukotrichia in vitiligo region | week12 after intervention
  average percentage reduction of leukotrichia in vitiligo region from baseline to week 12
NB-UVB dose | week12 after intervention
  Using the following Equation 1 : φ=E*T (E refers to irradiation intensity [mW/cm2] ; φ refers to irradiation dose [mJ/cm2]; T refers to irradiation time [sec]) to calculate the effective NB-UVB dose for patients at week 12

OTHER OUTCOMES:
number of participants with treatment-related events such as desquamation and dryness, erythema, and blister formation. | week12 after intervention
  safety assessment involved monitoring adverse events such as desquamation and dryness, erythema, and blister formation.

CONTACTS AND LOCATIONS:
Overall Officials: Lu Yan, Study Chair — The First Affiliated Hospital with Nanjing Medical University
Locations (1):
- The first Affiliated hospital with Nanjing medical university, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No